CLINICAL TRIAL: NCT06454682
Title: A Single-site, Single-arm, Open-label, IIT Clinical Study to Evaluate the Safety and Efficacy of a Single Intrathecal Injection of AAV-RJK002 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: An IIT Clinical Study to Evaluate the Safety and Efficacy of a Single Intrathecal Injection of RJK002 in Patients With ALS
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: RJK Biopharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJK-002-I
Record Dates: First submitted 2024-06-03; First posted 2024-06-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive a single intrathecal administration of investigational product. 9 subjects will be involved in 3 doses cohort from low to high: 3E13 vg/person, 6E13 vg/person, and 1.2E14 vg/person, 3 subjects for each cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RJK002 Intrathecal injection (Experimental)
  Interventions: Drug: RJK002 Intrathecal injection

INTERVENTIONS:
Drug: RJK002 Intrathecal injection — Eligible subjects will receive a single intrathecal administration of investigational product with dose 3E13 vg/person, 6E13 vg/person, and 1.2E14 vg/person sequentially.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of a single intrathecal injection of RJK002 in patients with Amyotrophic Lateral Sclerosis (ALS). The main questions it aims to answer are:

* The safety, tolerability, and preliminary efficacy of a single intrathecal injection of RJK002 in subjects with amyotrophic lateral sclerosis (ALS)
* The adeno-associated virus (AAV) viral load, changes of biomarkers in serum and cerebrospinal fluid (CSF), and electromyography (EMG) motor unit counts in subjects with ALS treated with a single intrathecal injection of RJK002.

Participants will receive a single intrathecal administration of investigational product and a systemic immunomodulatory regimen. There will be 3 cohorts: 3E13 vg/person (3 mL), 6E13vg/person (6 mL), and 1.2E14 vg/person (12 mL). 3 subjects will be enrolled in each dose cohort. The dose level will be escalated sequentially from low to high.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects who are ≥ 18 years of age at screening;
2. Patients with a diagnosis consistent with clinically or laboratory-supported possible, probable, or definite sporadic or familial ALSALS in accordance with Revised EI Escorial diagnostic criteria published by the World Federation of Neurology (WFN);
3. The duration of the disease from the first symptom (any ALS symptom) prior to the screening visit must be more than 6 months and less than 2 years (inclusive);
4. The Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) score ≥30 during the screening period, and the three respiratory scores (dyspnea, upright respiration, and respiratory insufficiency) must be full marks;
5. The forced vital capacity (FVC) of predicted during the screening period is ≥70% at screening;
6. Body mass index (BMI) greater than 18 kg/m2 at screening;
7. Subjects who had not taken riluzole, edaravone, or who had been on a stable dose for ≥30 days at screening and continue to take it during the study period (those who have stopped taking riluzole, edaravone for ≥ 30 days at screening may also be included, in the opinion of the Investigator);
8. Understand and comply with the trial procedure, voluntarily participate in and be willing to undergo genetic testing, and sign the informed consent (the informed consent is voluntarily signed by the subject or the subject's leagally authorized representative in the case that a subject is legally incapable of providing informed consent).

Exclusion Criteria:

1. Subjects with other neurological diseases similar to ALS that affect the evaluation of drug efficacy, such as cervical spondylotic myelopathy, syringomyelia, spinal cord and brain stem tumors, hirayama disease, multifocal motor neuropathy, multiple sclerosis, Guillain-Barre syndrome, Parkinson's disease and dementia;
2. Subjects who refuse to take food and medication by nasal feeding tube during the study period due to swallowing dysfunction;
3. Subjects with a history of spinal surgery within the last six months after the onset of ALS;
4. By cytological analysis at screening, the titer of anti-AAV9 neutralizing antibody was positive (>1:100);
5. AST, ALT, bilirubin, glutamyltransferase, or glutamate dehydrogenase >1.5 × ULN or serum creatinine (Scr) > ULN at screening;
6. Any medical instability deemed by the Investigator to be clinically significant, including but not limited to the presence of cardiovascular and cerebrovascular, hepatic or renal dysfunction, endocrine, psychiatric, or nervous system abnormalities that the investigator believes would interfere with the overall safety or efficacy of the study;
7. Subjects with history of convulsive seizures or epilepsy (excluding febrile convulsive seizures in childhood);
8. History of autoimmune diseases (excluding thyroid diseases), myelodysplastic or myeloproliferative diseases, leukemia or lymphoma, or severe scoliosis;
9. Subjects who are hospitalized for surgery, pulmonary events, or nutritional support within 2 months prior to the screening period or who planned to undergo hospitalization for major surgery during the study period;
10. Presence of contraindications to lumbar puncture (including, but not limited to, signs or symptoms of skin infection at the administration site and elevated intracranial pressure), receipt of any active intrathecal therapy, presence of implantable shunt tubes for draining cerebrospinal fluid (CSF), presence of implantable central nervous system (CNS) cannula, or any condition that interferes with CSF collection;
11. Screening for a record of attempted suicide in the six months prior to the screening visit, who indicated four or five categories of suicidal thoughts on the Columbia-Suicide Severity Rating Suicide Scale (C-SSRS) assessment, or who the Investigator judged to be at risk of suicide attempts;
12. Active infection requiring systemic antiviral or antibacterial therapy at any time between 4 weeks prior to the start of screening and dosing; Active but untreated viral or bacterial infection at any time between 4 weeks prior to the start of screening and dosing; Any febrile illness developed during the 2 weeks prior to the start of screening until treatment was given;
13. Suspect or have a history of alcohol or drug abuse;
14. Hepatitis B virus surface antigen, hepatitis C virus antibody, syphilis, or human immunodeficiency virus antibody positive at screening;
15. Pregnant or lactating female subjects, or subjects of childbearing potential (including heterosexual male subjects and their fertile female partners), who have pregnancy plans during the study period or do not want to use effective contraception during the study period;
16. Subjects who have been received any stem cell therapy or gene therapy prior to screening;
17. Subjects vaccinated within 2 weeks prior to screening or expected to be vaccinated during the study period;
18. Subjects with concomitant or ongoing immunosuppressive therapy within 90 days prior to IP administration;
19. Subjects who have participated in another clinical trial and received any investigational therapy within 3 months prior to screening;
20. Subjects who are deemed inappropriate by the investigator to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2031-08-02 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events (AEs)/serious adverse events (SAEs) | Each visit within 5 years after administration
Dose limiting toxicities (DLT) | 28 days after administration
  Measured as any drug-related serious adverse event that meet DLT standard. If a dose has less than 33% DLTs it will be considered tolerable.

SECONDARY OUTCOMES:
Change in the ALS Functional Rating Scale-revised (ALSFRSr) Score. | 28 days, 56 days, 84 days, 6 months, 12months, 18 months
  The ALSFRSr, a questionnaire-based scale assessing daily living function ranging from 48 (best score) to 0 (worst), was administered to the patient, or to a proxy if the patient could not communicate effectively. Decline was defined as ALSFRSr at baseline minus ALSFRSr at month 9. A positive value indicates worsening.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Some of data are planned to be shared on Nov 2025 and Nov 2026.